CLINICAL TRIAL: NCT00582101
Title: Family-Based HIV Prevention for Latinos
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Celia Lescano, Ph.D., Assistant Professor (Research), Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1K01MH078783-01 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections
Keywords: HIV; prevention; families; Latinos; communication; sexuality; monitoring; health promotion; HIV Prevention; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Communication; Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family-based HIV (Experimental)
  Interventions: Behavioral: Family-Based HIV Prevention for Latinos
- Family-based HP (Active Comparator)
  Interventions: Behavioral: General Health Promotion

INTERVENTIONS:
Behavioral: Family-Based HIV Prevention for Latinos — 7-hour one-day workshop with adolescents and parents in separate and joint sessions
  Other Names: Latino STYLE
  Arms: Family-based HIV
Behavioral: General Health Promotion — 7 hour one-day workshop on general health promotion topics
  Arms: Family-based HP

SUMMARY:
The proposed project will develop and test an HIV prevention intervention for Latino families. This study will:

1. Conduct a pilot "run-through" of an adapted family-based intervention with three cohorts (about 24 families) to determine the feasibility, acceptability, and appropriateness for the target population.
2. Revise the family-based HIV prevention intervention based on the results of the pilot "run-through" and structured exit interviews.
3. Recruit and randomize 100 families into the Latino family-based HIV prevention intervention or a general health promotion condition.
4. Estimate the effect size of the Latino family-based HIV prevention intervention from assessment of changes in HIV-related sexual behavior and attitudes and parental monitoring/supervision over 6 months.

Based on a thorough review of the literature, the following is anticipated:

1. The revised intervention will be feasible, acceptable, and appropriate for Latino families and will be enthusiastically received.
2. The family-based HIV prevention intervention will result in safer adolescent sexual behavior, greater change with regard to primary outcome measures of behavior (recent sexual activity, the number of unprotected sex acts, proportion of condom use, and intentions to use condoms), safer HIV-related attitudes, improved parent-child communication skills, and greater parental monitoring than the Latino families in the general health promotion condition.

DETAILED DESCRIPTION:
Latinos are disproportionately represented among those diagnosed with HIV and Latino adolescents are at risk for engaging in sexual behaviors that can lead to HIV. However, data regarding HIV prevention interventions for Latino adolescents, as distinct from other ethnic groups, have not been published to date. This K Award will conduct an initial study of a family-based intervention specifically for Latino families. With the support of a NIMH Minority Supplement Award, Dr. Lescano has adapted a family-based intervention from a multi-site trial for non-minority youth. Using a qualitative approach, Dr. Lescano has added to the intervention family context issues relevant to Latinos such as acculturation, religiosity, gender role and sexual socialization, parent-child communication, and monitoring practices. The initial phase of the K Award will be a run-through of the adapted family-based intervention with three cohorts (8 families per group) to further assess participant reaction and appropriateness. The intervention will then be revised based on feedback using structured exit interviews. Next, 100 Latino families with an adolescent between the ages of 13 and 18 will be randomized into either the family based HIV prevention intervention or a general health promotion (GHP) condition that focuses on healthy behaviors such as diet and exercise. Groups consist of 6 to 8 parent and youth dyads in a one-day, 7-hour workshop. Both interventions employ activities for youth and parents separately (e.g., focus on adolescent vulnerability) and parents and adolescents together. The project will estimate the effect size of the Latino Family-based HIV prevention intervention from assessment of changes in the adolescents' HIV-related sexual behavior and attitudes, gender and sexual socialization, parent-child communication, and parental monitoring. Measures will be completed at baseline and at 3 and 6 months post-intervention. The work done in this K Award will provide pilot data that will lead to submission of an R01 to determine the efficacy of the intervention, compared to a adolescent-only, skills-based HIV prevention group and a general health promotion group, in a larger sample of Latinos. An efficacious intervention is urgently needed for Latino communities.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent must be English-speaking and can converse in Spanish with parent
* Parent must be Spanish-speaking
* Adolescent and parent must be living together for at least 3 months prior to workshop
* Both parent and adolescent self-identify as being of Hispanic/Latino origin

Exclusion Criteria:

* Adolescent HIV positive
* Adolescent pregnant or intending to get pregnant
* Active psychosis

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2007-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Number (#) of unprotected sex acts | baseline, 3, and 6 months

SECONDARY OUTCOMES:
parent-child communication | baseline, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Celia M Lescano, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States